CLINICAL TRIAL: NCT04744246
Title: An Analysis of Muscle Activity During Load Carriage Activity in Army ROTC Cadets
Brief Title: Muscle Activity During Load Carriage in ROTC Cadets
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: North Dakota State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Screening
Other Study IDs: HE20208
Record Dates: First submitted 2020-05-21; First posted 2021-02-08 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Back Pain
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Without Load (Active Comparator): 5 kilometer walk with no load carried
  Interventions: Other: load carriage
- With Load (Experimental): 5 kilometer walk with load
  Interventions: Other: load carriage

INTERVENTIONS:
Other: load carriage — 35 pound load carried on the back

SUMMARY:
Army ROTC Cadets who are currently enrolled in Military Science courses will be asked to participate in this experimental research design. A total of 30 healthy cadets consisting of approximately 24 males and six females will be recruited, as this will provide an accurate representation of the overall Army demographics with 17% being female.

Paperwork: After providing consent, participants age and gender will be documented, and height and weight will be measured and documented. Participants will complete a modified version of the Modified Oswestry Low Back Pain Disability Questionnaire, which has been adjusted to be more specific to the military population. The questionnaire will be filled out indicating the cadet's current level of pain. They will then complete the same questionnaire indicating their pain within the last year.

Protocol: First, the skin will be prepared and surface electromyography (EMG) electrodes will be placed. Dynamic, surface EMG data will be obtained of the gluteus medius, gluteus maximus, erector spinae, rectus femoris, and biceps femoris muscles in accordance with SENIAM (Surface Electromyography for the Non-Invasive Assessment of Muscles) guidelines. Skin preparatation will consist of trimming hair if the skin surface at which the electrodes have to be placed is covered with hair. Next, the skin will be cleaned with alcohol. The skin will be allowed to dry prior to electrode placement. Lastly, skin will be abraded to reduce impedance. Following electrode application, participants will complete five minutes of light activity on a bike or treadmill for warm-up. Next, in order to normalize the data, manual muscle tests will be performed for each of the six muscles being test. Then, participants will walk at a speed of four miles per hour for 10 seconds as a dynamic measurement for normalizing the data.

After completion of the two normalization protocols, participants will complete a five kilometer (3.1 mile) walk on a treadmill at a speed of three miles per hour, with and without a 35 lb. load carried in a traditional rucksack. The load conditions will be randomized and counterbalanced in order to mitigate effects of fatigue, and the conditions will be performed in two separate sessions (separated by 24-48 hours).

ELIGIBILITY:
Inclusion Criteria:

* current enrollment in military science courses and member of Army ROTC

Exclusion Criteria:

* current musculoskeletal injuries

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-09-07 (Actual); Primary Completion 2020-10-29 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
EMG change over time with Load carriage | 2 days
  muscle activation of rectus femoris, gluteus medius, gluteus maximus, biceps femoris, rectus abdominis, and erector spinae with a 35 lb load
EMG change over time without load | 2 days
  muscle activation of rectus femoris, gluteus medius, gluteus maximus, biceps femoris, rectus abdominis, and erector spinae without a 35 lb load
Modified version of Modified Oswestry Disability Index Current Pain | 1 day
  answers to back pain questionnaire for current level of pain
Modified version of Modified Oswestry Disability Index Pain in Last Year | 1 day
  answers to back pain questionnaire for any pain within the last year

CONTACTS AND LOCATIONS:
Locations (1):
- North Dakota State University, Fargo, North Dakota, United States

IPD SHARING:
Plan to Share IPD: No